CLINICAL TRIAL: NCT04010682
Title: Late Pregnancy Sample Collection Study
Status: Completed | Type: Observational
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PROTOCOL-1095
Record Dates: First submitted 2019-06-19; First posted 2019-07-08 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Daily urine samples collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: urine sample collection — no drug/devise intervention. sample collection study only

SUMMARY:
This study will obtain daily urine samples from pregnant volunteers, from 36 weeks pregnant until birth. All urine samples will be stored and used for research or product validation purposes.

The study will also gather information from volunteers regarding a woman's health during her pregnancy.

DETAILED DESCRIPTION:
This study will obtain daily urine samples from pregnant volunteers, from 36 weeks pregnant until birth. It is anticipated 20-40 pregnant women will be recruited to the study.

Urine samples will be delivered to SPD either via post, or by hand and form part of the SPD BioBank. All urine samples will be stored and used for research or product validation purposes.

The study will also gather information from volunteers regarding a woman's health during her pregnancy, including any bleeding, discharge, discomfort, contractions/ Braxton Hicks via the use of a daily diary.

Pregnancy outcome details including labour specifics and birth outcomes such as birth date, weight, and sex of the baby will be obtained 4-6 weeks after the volunteer has given birth via email correspondence between the volunteer and study co-ordinator.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant female in 3rd trimester of pregnancy

Exclusion Criteria:

* Prescribed bed-rest during third trimester or any other pregnancy
* complication that would affect the ability to participate in the study
* more than 38 weeks pregnant
* Have a planned caesarean section

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: healthy pregnant volunteers
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
late pregnancy urine samples | 4 weeks
  Number of volunteers providing daily urine samples from 36 weeks pregnant until birth.

SECONDARY OUTCOMES:
pregnancy complications | 6 weeks
  Number of participants reporting pregnancy complications from week 36 of pregnancy until birth
Live birth | 6 weeks
  number of study participants who's pregnancy resulted in a live birth
Spontaneous vaginal delivery | 6 weeks
  number of study participants who's pregnancy resulted in a spontaneous vaginal delivery
weight of baby | 6 weeks
  weight of baby in pounds and ounces or kilograms
multiple births | 6 weeks
  number of pregnancies resulting in single baby, twins or triplets.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Johnson, Study Director — SPD Development company Ltd.
Locations (1):
- SPD Development Company Ltd, Bedford, Bedfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No